CLINICAL TRIAL: NCT00513786
Title: A Phase II Study of Carboplatin/Paclitaxel/Bevacizumab in the Treatment of Advanced Stage Endometrial Carcinoma
Brief Title: Evaluation of Carboplatin/Paclitaxel/Bevacizumab in the Treatment of Advanced Stage Endometrial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David O'Malley (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David O'Malley, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06133; NCI-2012-01229 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Advanced Stage Endometrial Cancer; Stage 3 or 4 endometrial cancer; Cancer treatment; gyn cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- carboplatin/paclitaxel with bevacizumab (Experimental): A regimen of Carboplatin and paclitaxel combined with bevacizumab given every 21 days in patients with advanced stage endometrial cancer for a maximum of 6 cycles.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: bevacizumab

INTERVENTIONS:
Drug: Carboplatin — AUC (area under curve) 5 Intervenous (IV) over 30 minutes given every 21 days for a maximum of 6 cycles.
  Other Names: Paraplatin; CBDCA
Drug: Paclitaxel — 175 mg/m2 over 3 hours given every 21 days for a maximum of 6 cycles.
  Other Names: Onxol; Taxol
Drug: bevacizumab — 15 mg/kg intervenous (IV) given every 21 days for a maximum of 6 cycles.
  Other Names: Avastin

SUMMARY:
Purpose of this study is to determine the effectiveness of the drug combination carboplatin, paclitaxel, and bevacizumab(Avastin) in patients with advanced stage endometrial carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness, safety, and tolerability of the drug combination carboplatin, paclitaxel, and bevacizumab(Avastin) in patients with advanced stage endometrial carcinoma. This is a phase II,open label,single center study. Patients will receive carboplatin, paclitaxel, and bevacizumab in an outpatient center by intravenous administration. The primary objectives is to study the progression free survival at 24 months after initiation of treatment and to determine the toxicity profile of the drug combinations. The secondary objectives are to estimate the overall survival and tumor response for this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Stage Endometrial Cancer (Stage 3 or 4)
* Any Histology including clear cell, and serous papillary carcinomas
* surgery must have had hysterectomy and bilateral salpingo-oophorectomy
* chemotherapy initiated 12 weeks after surgery
* sign informed consent
* Adequate End-organ function
* GOG (Gynecologic Oncology Group)Performance Status 0,1,2
* Patients must be 18 years or older
* Patients may have received radiation for the treatment of endometrial cancer.
* Patients may have measurable or non-measurable disease.

Exclusion Criteria:

* Patient with concomitant malignancy other than non-melanoma skin cancer
* Patients with prior malignancy who have been disease free for 5 years.
* Patients with serious uncontrolled infection, angina or serious peripheral neuropathy.
* Patients whose circumstances will not permit study completion or adequate follow up
* Patients who have received prior cytotoxic chemotherapy for treatment of endometrial cancer including chemotherapy used for radiation sensitization.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O'Malley, MD, Principal Investigator — The Ohio State University Division of Gyn Oncology
Locations (1):
- The Ohio State University-Division of Gyn Oncology, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Patients With Progression Free Survival (PFS)
Description: Progressive Disease (PD) is defined at least a 20% increase in the sum of the longest dimension of target lesions, taking as reference the smallest sum of the longest dimension recorded since the treatment start or the appearance of one or more new lesions.
Time Frame: up to 57 months
Measure: Median (Full Range); unit: months
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
Number analyzed (Participants) | 38
months | 26 [2 to 57]

2. Secondary Outcome: To Estimate Overall Survival
Time Frame: up to 24 months
Population: Two participants did not complete all 24 months of follow-up and are were not analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
Number analyzed (Participants) | 36
percentage of participants | 69.4

3. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability.
Description: Toxicities will be assessed by using the NCI Common Toxicity Criteria for Adverse Events 3.0
Time Frame: up to 24 months
Measure: Number; unit: participants
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
Number analyzed (Participants) | 38
participants
  Patients with Adverse Event | 38
  Patients with Serious Adverse Event | 4

4. Secondary Outcome: Objective Tumor Response Using Modified RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
Description: Tumor response will be evaluated using modified RECIST criteria with the following definitions. Complete Response (CR) is disappearance of gross evidence of disease with confirmation at least 4 weeks later. Partial Response (PR) is a 30% or greater reduction in measurement of longest dimension of each lesion with confirmation at least 4 weeks later. Progressive Disease (PD) is at least a 20% increase in the sum of the longest dimension of target lesions, taking as reference the smallest sum of the longest dimension recorded since the treatment start or the appearance of one or more new lesions. Stable Disease (SD) is any condition not meeting the other criteria for CR, PR or PD.
Time Frame: Up to 24 months
Population: Two patients did not complete all 24 months of follow up and were not analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
Number analyzed (Participants) | 36
Participants
  Complete Response | 19
  Partial Response | 2
  Stable Disease | 7
  Progressive Disease | 1
  Unable to Determine | 3
  Zero Measurable Disease | 4

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Carboplatin/Paclitaxel With Bevacizumab
All-Cause Mortality (participants affected / at risk) | 11/38
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel With Bevacizumab (N=38)
Evisceration- fascia dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Evisceration- vaginal dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin/Paclitaxel With Bevacizumab (N=38)
Abnormal Creatinine (Investigations) | 12 (37)
Allergy/Immunology (Immune system disorders) | 2 (5)
Neutrophils/granulocytes (Investigations) | 12 (35)
Auditory/Hearing- other (Ear and labyrinth disorders) | 2 (2)
Cardiovascular Disorders (Cardiac disorders) | 15 (37)
Coagulation (Investigations) | 3 (4)
Constaipation (Gastrointestinal disorders) | 14 (44)
Dermatology disorders (Skin and subcutaneous tissue disorders) | 12 (39)
Diarrhea (Gastrointestinal disorders) | 8 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Increased Liver Enzymes (Investigations) | 5 (11)
Fatigue (General disorders) | 24 (67)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3)
Hemoglobin (Blood and lymphatic system disorders) | 12 (44)
Hemorrhage (Gastrointestinal disorders) | 3 (7)
Infection clinically documented (Infections and infestations) | 5 (7)
Lymphatics (Blood and lymphatic system disorders) | 4 (5)
Mucositis/stomatis (Gastrointestinal disorders) | 6 (16)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 17 (42)
Ocular/visual (Eye disorders) | 3 (5)
Other constitutional toxicity (General disorders) | 5 (20)
Other GI toxicity (Gastrointestinal disorders) | 8 (27)
Other infection toxicity (Infections and infestations) | 5 (11)
Other metabolic/lab toxicity (Investigations) | 11 (22)
Other neurologic toxicity (Nervous system disorders) | 7 (20)
Other pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (18)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (5)
Depression (Psychiatric disorders) | 3 (4)
Insomnia (Psychiatric disorders) | 12 (21)
Mood alteration (Psychiatric disorders) | 6 (8)
Taste alteration (Nervous system disorders) | 2 (2)
Pain, not specified (General disorders) | 19 (46)
Sensory neuropathy (Nervous system disorders) | 12 (39)
Platelet count decreased (Investigations) | 4 (14)
Vomiting (Gastrointestinal disorders) | 5 (9)
White blood cell decreased (Investigations) | 17 (50)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-01-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT00513786/Prot_SAP_000.pdf